CLINICAL TRIAL: NCT04424381
Title: Pharmacokinetics and Bioequivalence of Generic and Branded Rivaroxaban Tablet in Healthy Chinese Volunteers Under Fasting and Fed Conditions
Brief Title: Pharmacokinetics and Bioequivalence of Rivaroxaban Tablet in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: QL-YK4-012-001
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Healthy Subjects
Keywords: rivaroxaban; pharmacokinetics; bioequivalence
MeSH Terms: interventions — Rivaroxaban; Tablets

STUDY DESIGN:
Intervention Model Description: The study was designed as a four-period complete and replicate crossover
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rivaroxaban 20 MG Oral Tablet [Xarelto] (Active Comparator): rivaroxaban oral tablet [Xarelto] at a single oral dose of 20 mg
  Interventions: Drug: Rivaroxaban 20 MG Oral Tablet
- Rivaroxaban 20 MG Oral Tablet (Experimental): rivaroxaban oral tablet at a single oral dose of 20 mg
  Interventions: Drug: Rivaroxaban 20 MG Oral Tablet [Xarelto]

INTERVENTIONS:
Drug: Rivaroxaban 20 MG Oral Tablet [Xarelto] — The subjects randomly received single oral administration of Rivaroxaban 20 MG Oral Tablet [Xarelto].
  Arms: Rivaroxaban 20 MG Oral Tablet
Drug: Rivaroxaban 20 MG Oral Tablet — The subjects randomly received single oral administration of Rivaroxaban 20 MG Oral Tablet.
  Arms: Rivaroxaban 20 MG Oral Tablet [Xarelto]

SUMMARY:
The study was designed as a single-site, randomized, open-label, four-period complete and replicate crossover. A single oral dose of 20 mg rivaroxaban tablet (test) and Xarelto®(reference) was given to the 72 healthy Chinese adult volunteers, with 36 in a fasting state and 36 receiving a high-fat diet.

DETAILED DESCRIPTION:
Subjects were randomized into two treatment sequence groups: Sequence 1 = TRTR and Sequence 2 = RTRT, and each study period was separated by a 7 days washout period. After an overnight fast for at least 10 h, the subjects received a single oral dose of the R or T formulation of rivaroxaban tablets (20 mg) with 240 mL of water in a seated position. A total of 19 blood samples were collected at 0 (within 60 min prior to dosing) and 0.25,0.5, 1.0, 1.5, 2.0, 2.5,3.0,3.5, 4.0, 4.5,5.0, 5.5,6.0, 8.0, 12.0, 24.0, 36.0 ,and 48.0 hours after dosing.Blood samples were collected in a vacuum blood tube containing sodium heparin, gently mixed, and stored on ice-water mixture until sample processing and then centrifuged at 2000g at 2-8°C for 10 min.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 18 and above.
* The body mass index is in the range of 19.0-26.0 kg/m2 (including the critical value). The weight of male is not less than 50.0 kg, and that of female is not less than 45.0 kg.
* The following examination show that the indicators are normal or abnormal without clinical significance. The examination including: Vital signs, physical examination, blood routine, blood biochemistry, urinalysis, pregnancy test for female, serological tests for hepatitis B virus, hepatitis C virus, human immunodeficiency virus (HIV), and syphilis virus, 12 lead ECG, breath test for alcohol, drug abuse test.
* The subjects have no family planning within 3 months and could select contraceptive method.Before the study, all subjects
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.

Exclusion Criteria:

* Being allergy to the study medications, smoking, alcohol abuse.
* Participation in another clinical trial within 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 94 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 94 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 94 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 94 days
  Collection of adverse events
Incidence of abnormal blood pressure | 94 days
  Monitor the blood pressure
Incidence of abnormal temperature | 94 days
  Monitor the temperature
Incidence of abnormal pulse | 94 days
  Monitor the pulse
Incidence of abnormal electrocardiogram waveform | 94 days
  Electrocardiogram inspection

CONTACTS AND LOCATIONS:
Overall Officials: yu Cao, Principal Investigator — the study director of phase I clinical research center
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: No
All the technical achievements and outcomes of this trial are owned by Qilu Pharmaceutical Co., Ltd. and the research center. The research center can not publish any academic papers without the consent of the sponsor